CLINICAL TRIAL: NCT06603883
Title: Efficacy of Fecal Microbiota Transplantation in Critically Ill ICU Patients With Gastrointestinal Dysfunction-induced Enteral Nutrition Intolerance: a Single-center, Non-blind, Randomized Controlled Study
Brief Title: Efficacy of Fecal Microbiota Transplantation in ICU Patients With Gastrointestinal Dysfunction-induced Enteral Nutrition Intolerance
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiancheng Zhang, Prof. Jiancheng Zhang, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJC202408
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Dysfunction-induced Enteral Nutrition Intolerance
Keywords: FMT; Gastrointestinal dysfunction; ICU
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Receive ICU standard treatment.
- FMT intervention Group (Experimental): In addition to ICU standard treatment, 50ml commercial intestinal bacterial suspension was administered via a naso-jejunal tube to the jejunum from 11:00 to 13:00 every day for 3 consecutive days.
  Interventions: Biological: Fecal microbiota transplantation (FMT) by nasal jejunal tube

INTERVENTIONS:
Biological: Fecal microbiota transplantation (FMT) by nasal jejunal tube — FMT was administered via a naso-jejunal tube to inject 50ml commercial intestinal bacterial suspension into the jejunum.
  Arms: FMT intervention Group

SUMMARY:
Considering that intestinal microbiota plays a crucial role in intestinal function, fecal microbiota transplantation (FMT) may provide a new therapeutic strategy for the treatment of intestinal nutrition intolerance in critically ill ICU patients. The purpose of this study was to investigate the effects of FMT on the recovery of gastrointestinal dysfunction-induced enteral nutrition intolerance in critically ill patients admitted to ICU, and observe the effects on gastrointestinal barrier function, as well as the effects on length of stay in ICU, ICU mortality, in-hospital mortality, and 28-day mortality.

DETAILED DESCRIPTION:
Patients in the intensive care unit (ICU) are often at risk for gastrointestinal dysfunction and malnutrition. Gastrointestinal dysfunction is associated with poorer clinical outcomes, including longer mechanical ventilation, longer ICU stay, and increased 90-day mortality. Due to the influence of primary severe diseases and the use of proton pump inhibitors (PPI) and antibiotics, ICU patients with severe illness may have severe disturbance of intestinal flora, impairment of intestinal barrier function, high incidence of gastrointestinal dysfunction-induced enteral nutrition intolerance, and severe intestinal systemic inflammation and organ function injury. Considering that intestinal microbiota plays a crucial role in intestinal function, fecal microbiota transplantation (FMT) may provide a new therapeutic strategy for the treatment of gastrointestinal dysfunction-induced enteral nutrition intolerance in critically ill ICU patients. The project plans through nasal jejunal tube way to give FMT, to investigate its effect on the recovery of gastrointestinal dysfunction-induced enteral nutrition intolerance in severe patients admitted to ICU, and to observe its effect on gastrointestinal barrier function.

ELIGIBILITY:
Inclusion criteria:

1. 8 ≤ age ≤ 70 years old, any nationality, any gender;
2. Female patients have no potential fertility (i.e., no physical ability to conceive, including women who have been menopausal for 2 years) or no pregnancy plan;
3. Patients who have been in the ICU for at least 24 hours;
4. Patients with an expected ICU stay of at least 7 days;
5. Non-acute patients with at least one manifestation of gastrointestinal dysfunction leading to enteral nutrition intolerance;
6. Patients can cooperate or passively complete the relevant examination and complete the follow-up;
7. Informed consent is documented by means of a written, signed and dated informed consent form.

Exclusion Criteria:

1. Severe systemic infection, in early recovery period, hemodynamic instability or tissue hypoperfusion, severe imbalances in water and electrolyte status;
2. Patients who are considered by clinicians to be at high risk of death within 5 days, or who are subject to restricted treatment decisions;
3. Severe damage of intestinal barrier such as active massive bleeding and perforation of digestive tract;
4. Patients who cannot tolerate 50% of caloric calorie requirements with enteral nutrition due to severe diarrhea, significant fibrous intestinal stenosis, severe gastrointestinal bleeding, high-flow intestinal fistula and other reasons;
5. Nasal jejunal tube cannot be placed;
6. Planned or recent abdominal surgery (within 14 days);
7. Currently diagnosed with fulminant colitis or toxic megacolon;
8. Neutropenia (neutrophil count < 1500 /µL);
9. Patients with congenital or acquired immune deficiency;
10. Malignant hematologic diseases, such as lymphoma;
11. Autoimmune diseases;
12. Patients who have recently received high-risk immunosuppressive or cytotoxic drugs, such as rituximab, doxorubicin, or medium-high dose of steroid hormones (20mg/day or higher) for more than 4 weeks;
13. Pregnant or lactating women;
14. Participating in other clinical studies as a participant at the time of enrollment or within 3 months before inclusion;
15. Informed consent can not be obtained.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-19 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of the effective improvement of enteral nutrition intolerance | 24, 48, 72 and 96 hours after first FMT.
  Change of intestinal nutrition intolerance.

SECONDARY OUTCOMES:
Changes of intestinal microbiota and its metabolites | -48, 72 and 96 hours after first FMT.
  Rectal swab was taken and analysed by 16S rRNA gene sequencing and metabolomics.
Intestinal barrier function | -24, 0, 24, 48, 72 and 96 hours after first FMT.
  2ml of peripheral venous blood was collected for the measurement of serum lipopolysaccharide (LPS), diamine oxidase (DAO), and D-lactic acid.
Acute gastrointestinal injury (AGI) score | -48, -24, 0, 24, 48, 72 and 96 hours after first FMT.
  Acute gastrointestinal injury (AGI) score is quoted from the "Expert consensus on enteral nutrition for gastrointestinal dysfunction in critically ill patients (2021 edition)". AGI can be divided into Ⅰ, Ⅱ, Ⅲ and Ⅳ grades, and the higher the grade, the more serious the gastrointestinal dysfunction.
Acute Physiology and Chronic Health Evaluation (APACHE) Ⅱ score | -48, -24, 0, 24, 48, 72 and 96 hours after first FMT.
  Acute Physiology and Chronic Health Evaluation (APACHE) Ⅱ score is a scoring system used to assess the severity of critically ill patients. APACHE II score ranges from 0 to 71. The higher the score, the greater the severity and the poorer the prognosis.
C-reactive protein (CRP) and procalcitonin (PCT) | -48, -24, 0, 24, 48, 72 and 96 hours after first FMT.
  2ml of peripheral venous blood was collected for the measurement of CRP and PCT.
Peripheral blood cytokines and lymphocyte subsets | -24 and 72 hours after inclusion.
  2ml of peripheral venous blood was collected for the measurement of the levels of cytokines and the absolute number of lymphocyte subsets.
ICU mortality | From date of randomization until the date of discharge from the ICU or date of death from any cause during ICU stay, whichever came first, assessed up to 6 weeks
  Mortality rate of patients in each group during their stay in the ICU.
In-hospital mortality | From date of randomization until the date of discharge from the hospital or date of death from any cause during hospitalization, whichever came first, assessed up to 6 weeks
  Mortality rate of patients in each group during hospitalization.
28-day mortality | 28 days after inclusion.
  Mortality rate of patients in each group within 28 days after inclusion.
90-day mortality | 90 days after inclusion.
  Mortality rate of patients in each group within 90 days after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jiancheng Zhang, Dr., Principal Investigator — Wuhan Union Hospial
Locations (2):
- China (2):
  - Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No